CLINICAL TRIAL: NCT01096953
Title: A Randomized Exploratory Study of Telepsychiatry Outcomes in Rural Youth
Brief Title: Telepsychiatry in Rural Youth
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not human subject research
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1R21MH079984-01 (NIH)
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; attention deficit
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telepsychiatry (Active Comparator): Psychiatry provided over telehealth network
  Interventions: Behavioral: Mental health care implemented by telepsychiatry; Behavioral: Face-to-face care
- Face-to-face care (Active Comparator): Psychiatry provided in person
  Interventions: Behavioral: Face-to-face care

INTERVENTIONS:
Behavioral: Mental health care implemented by telepsychiatry — Care of 6-17 year-olds with ADHD
  Arms: Telepsychiatry
Behavioral: Face-to-face care — Psychiatry provided for treatment of ADHD face-to-face in office

SUMMARY:
1. It is difficult to offer kids who live in rural areas good psychiatric care. There are only about 7000 psychiatrists for kids (pediatric psychiatrists) in the entire country. When adding nurse practitioners who specialize in mental health care for children, there still are not enough for everyone who needs care. This means either delays in treatment or no treatment at all by these important specialists. The purpose of this study is to explore how the investigators might offer psychiatric care to kids who live in rural areas through the use of telepsychiatry (TP), specifically those with attention deficit/hyperactivity disorder (ADHD).

   TP is a way for a physician to talk to someone in a remote area using a computer. The investigators will split the subjects into two study groups. As subjects are identified, they will be assigned a screening number according to a randomization table. The investigators will use TP for one group and face-to-face (F2F) care for the other group. The computer will allow the physician to look at and talk with the child and their parent(s). The investigators would like to know if TP is as good as, or nearly as good as F2F care, so the only difference in treatment approach between the two groups will be whether the subject is receiving treatment through TP or F2F care. Treatment is standardized using a flow chart called the Children's Medication Algorithm Project (CMAP) algorithm. The CMAP algorithm is a guideline established by a large number of experts who have agreed on the best approach to treatment based on scientific evidence. If TP proves as good as F2F care, it would help many parents and their children who do not live in or near a large city.
2. The investigators will find study subjects when parents seek care at clinics in rural Oregon. The physicians in those locations will be aware of the study and will tell us when they think someone needs specialized mental health professional (either a pediatric psychiatrist or nurse practitioner with extensive experience in pediatric mental health). The investigators will make sure that ADHD is the right diagnosis using special exams that have been well-tested to show that they are reliable.
3. The first visit-the intake visit-will probably take about an hour. At that visit, mental health professional will determine whether or not the patient is a candidate for the study. If the patient agrees, they will be asked to sign consent and child assent. The parent and child will then be given an exam that will confirm the diagnosis of ADHD. If confirmed, subjects will then learn if they have been assigned to the TP group or the F2F group and will be assigned to the treating mental health professional. In addition to the DISC, after consent the parent will be given several study instruments to take home with them. They will take about an hour altogether to complete.

   The first visit with the treating mental health professional will take about one hour and the three following visits will take about 30 minutes each. These visits will be about six weeks apart. At the third follow-up visit-the final visit-the parents will be again asked to complete the instruments they completed after consent and will be asked to complete a brief questionnaire that will give them the opportunity to describe their satisfaction or dissatisfaction with the treatment and care they received.

   Teachers will be asked to complete the Conner's 10-Item Global Index for the subject twice over the course of the study. The parent of the subject will present the scale to the teacher and retrieve the scale in a sealed envelope to return to the clinic.
4. The diagnosis for ADHD will be made using an exam called the Diagnostic Interview Schedule for Children Version IV (DISC IV). This is a 90-minute exam that is done with a computer that helps you know what questions to ask and helps record the responses. The parents will also be asked to complete a few instruments and surveys that help us understand how well treatment is working. The investigators expect these exams to take about half an hour to complete. They contain questions about the subject's behavior and are completed by parents, except one brief instrument that the investigators will ask and teachers to complete before each follow-up visit. These instruments take about 10 minutes each to complete.
5. This is an initial "pilot" study, so the information collected will mainly offer a better understanding of whether or not a larger study is possible. The investigators will look at how many subjects stayed in the study or dropped out and when they dropped out. The investigators will also look at the exams, scoring them to help us understand if those who were part of the TP group did as well, or nearly as well, as those in the F2F group.

ELIGIBILITY:
Inclusion Criteria:

Inclusions:

The study will include children with co-occurring psychiatric conditions because of high comorbidity rates in ADHD. Comorbidity is present in as many as two-thirds of children with ADHD, including up to 50% for other disruptive disorders, 15%-20% for mood disorders, 20% to 25% for anxiety disorders, and 15-20% for learning disorders (Dulcan et al., 1997). Thus, with inclusion of children with comorbidity, the findings will have greater generalizability. Additionally, the comorbid children and adolescents are often too complex for primary care treatment and need child psychiatric services. The study will include:

1. Learning disorders, such as Mathematics Disorder, Reading Disorder, and Disorders of Written Expression.
2. Other disruptive disorders, such as (oppositional Oppositional defiant Defiant disorder Disorder and conduct Conduct disorder.)
3. Unipolar mood disorders, including Major Depressive Disorder and Dysthymic Disorder
4. Anxiety disorders hat coexist with ADHD, anxiety, and
5. Post traumatic stress disorder (PTSD).
6. Non-rapid cycling bipolar disorder stable on medications

Exclusions:

As in Pliszka et al.'s (2003) study of the CMAP ADHD treatment algorithm, only conditions that would prevent treatment for the primary disorder from being effective will be excluded. The study will not include subjects with:

Exclusion Criteria:

1. Rapid cycling bipolar disorder
2. A history of psychosis of any etiology. (Exceptions may include temporary medically or pharmacologically induced delirium.)
3. Medically impairing eating disorders,
4. Substance abuse within the past year or "active substance use"
5. Mental retardation (IQ < 70)
6. Autism spectrum disorders.

Children and families who are not English speaking will not be included in the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Equivalence | 4/15/2010-9/15/2011
  The number of visits completed by subjects assigned to the telepsychiatry arm will be "equivalent" to the number completed by subjects assigned to the face-to-face arm. Follow-up retention is directly associated with psychiatric outcomes and it is possible that telehealth might be seen by participants as somewhat impersonal. The implication is that retention will be reduced in the telepsychiatry group compared to the face-to-face arm. Retention will be defined as visits from baseline to either drop-out or completion of the four-month f/u study period. Visits occur at monthly intervals.

SECONDARY OUTCOMES:
Non-inferiority | 4/15/2010-9/15/2011
  Telehealth will be non-inferior to face-to-face services with regard to the change in the inattention component of attention-deficit / hyperactivity disorder symptoms measured at baseline and at the end of the four-month intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy C Winters, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Douglas County Health & Social Services, Roseburg, Oregon, United States